CLINICAL TRIAL: NCT00181272
Title: Macrolides to Prevent Exacerbations of Asthma and Chronic Obstructive Pulmonary Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Principal Investigator moved institutions
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Jerry A. Krishnan, Associate Professor, Johns Hopkins University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 05-02-17-01
Record Dates: First submitted 2005-09-15; First posted 2005-09-16 (Estimated); Last update posted 2013-05-13 (Estimated); Status verified 2013-05

CONDITIONS: Asthma; Chronic Obstructive Pulmonary Disease
Keywords: chronic obstructive pulmonary disease (COPD); undifferentiated asthma/COPD
MeSH Terms: conditions — Asthma; Pulmonary Disease, Chronic Obstructive | interventions — Azithromycin

INTERVENTIONS:
Drug: azithromycin

SUMMARY:
The purpose of this study is to determine whether macrolide therapy is effective in treating patients hospitalized with asthma exacerbations or chronic obstructive pulmonary disease (COPD)exacerbations. We hypothesize that compared to placebo, maintenance therapy with macrolides, when added to usual care, a) improves respiratory symptoms, b) improves quality of life, c) reduces airway inflammation, d) reduces airflow obstruction, and e) decreases the rate of re-exacerbations.

DETAILED DESCRIPTION:
Asthma and chronic obstructive pulmonary disease (COPD) are the two most common obstructive lung diseases. Chronic airway inflammation and episodic worsening of respiratory symptoms and airflow obstruction (exacerbations) occur in asthma and COPD. Despite major advances in the development of therapies for these respiratory disorders, asthma and COPD exacerbations are common and result in substantial morbidity and mortality. Moreover, patients hospitalized for asthma or COPD exacerbations are at high risk for near fatal and fatal re-exacerbations after discharge home. These observations highlight the need for novel therapies to prevent asthma and COPD exacerbations. The role of macrolide antibiotics (e.g., azithromycin, clarithromycin, erythromycin) in treating bacterial infections is well established. Recent pre-clinical evidence also suggests that macrolides may posses distinct anti-inflammatory properties and even anti-viral properties. These exciting observations have led to research evaluating the use of maintenance therapy with macrolides in patients with asthma and COPD. Small studies in clinically stable asthma or COPD suggest that maintenance macrolide therapy (e.g., use for 6 weeks), when added to usual care, may attenuate airway inflammation, reduce respiratory symptoms, and improve lung function. However, there are no studies that have evaluated the potential benefits of initiating maintenance macrolide therapy during asthma or COPD exacerbations. We hypothesize that initiating maintenance macrolide therapy in hospitalized patients with asthma or COPD exacerbations will, when added to usual medical care, accelerate the improvement in airflow obstruction, respiratory symptoms, and quality of life and reduce the risk of re-exacerbations after discharge home. The objective of this pilot study is to evaluate the feasibility of the study protocol (recruitment, retention, and adherence to study procedures and medications), as well as collect preliminary data about the proportion of exacerbations due to bacterial or viral infections and estimate potential effect sizes for clinically important outcomes (respiratory symptoms, quality of life, airflow obstruction, airway inflammation, and rate of re-exacerbations). To achieve these objectives, we propose a 48 week randomized, double-blind, placebo-controlled crossover clinical trial (24 weeks azithromycin, 24 weeks placebo) in adults hospitalized for asthma or COPD exacerbations to the Johns Hopkins Hospital or Johns Hopkins Bayview Medical Center.

ELIGIBILITY:
Inclusion Criteria:

* Physician-diagnosis of asthma, COPD exacerbation, or undifferentiated asthma/COPD exacerbation
* Admitted to the inpatient medical service at Johns Hopkins Hospital or Johns Hopkins Bayview Medical Center
* Evidence of airflow obstruction on spirometry (FEV1/FVC<70%)
* Age 18 years or older

Exclusion Criteria:

* History of allergy or other contraindication to macrolides (azithromycin, erythromycin, clarithromycin)
* Treatment with any macrolide in the 4 weeks prior to study entry
* Elevated AST or ALT (2 or more times the upper limit of normal) on current admission
* Elevated alkaline phosphatase (>1.25 times the upper limit of normal) on current admission
* Elevated total serum bilirubin (more than upper limit of normal) on current admission
* Previous participation in this study
* Patients prescribed digoxin (azithromycin may increase digoxin levels)
* Patients prescribed warfarin (azithromycin may increase INR in patients on warfarin)
* Patients prescribed pimozide (azithromycin may increase risk of arrhythmias)
* Patient unable to provide consent (e.g., language difficulty or history of dementia)
* Patient to be discharged to a location other than home (e.g., other hospital, long-term care facility)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2005-09; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
The effect of azithromycin on the rate of exacerbations for asthma or COPD exacerbations after hospital discharge

SECONDARY OUTCOMES:
changes in airflow obstruction (FEV1% predicted)
serum biomarkers of airway inflammation (IL-1beta, IL-5, IL-6, IL-8, IL-10, RANTES, IFN-gamma, TNF-alpha, and hs-CRP)
respiratory markers of inflammation (EBC measurements - pH)
symptom/quality of life measures

CONTACTS AND LOCATIONS:
Overall Officials: Jerry A Krishnan, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States